CLINICAL TRIAL: NCT02301832
Title: Reliability of Sensor Spacing for Near Infrared Spectroscopy in Traumatic Tibia Fractures: An Observational Study
Brief Title: Reliability of Sensor Spacing for NIRS in Traumatic Tibia Fractures
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William Reisman, William Reisman MD, Emory University
Other Study IDs: IRB00075483
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Orthopedic Disorders; Tibial Fractures
Keywords: acute compartment swelling (ACS); near-infrared spectroscopy (NIRS)
MeSH Terms: conditions — Musculoskeletal Diseases; Tibial Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study intended to evaluate a non-invasive device that uses light to measure the amount of oxygen in the muscles of injured and non-injured legs in specific situations. The name of this technology is NIRS (near-infrared spectroscopy). The goal of this study is to collect the information necessary to understand the use of the NIRS monitoring system to diagnose and direct treatment decisions in case of complications sometimes experienced in traumatic tibia fracture, such as excessive swelling called acute compartment syndrome (ACS).

DETAILED DESCRIPTION:
This study seeks to further develop the use of NIRS technology in the diagnosis of acute compartment syndrome. NIRS values normally increase in traumatized legs compared to the contralateral uninjured leg or forearm, indicative of a hyperemic response. The investigators hopes to build upon the current knowledge and verify the ability to accurately detect ACS using two easily identified and accessible leg compartments, the anterior and superficial posterior utilizing the Nonin 7600 oximeter with the Sensor Model 8004CV. Additionally, since this device was originally designed with brain tissue in mind, the NIRS device will collect vital engineering data that will be used to validate the algorithm used to produce the oxygenation values in injured muscle tissue.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral leg injury
* Enrolled within 48 hours of injury
* Subjects with 'severe' leg injuries presenting at trauma center that meet at least one of the following from each group below:

Anatomic location:

* Tibia/Fibula shaft fracture
* Tibial plateau fracture (Schatzker III-VI)

High Energy Mechanism of Injury:

* Fall from >8 foot height
* Motor vehicle collision (> 15 mph)
* Motor vehicle versus pedestrian accident
* High velocity gunshot wound
* Crush injury
* Sport/recreation

Exclusion Criteria:

* Application of NIRS monitoring would be an impediment to care
* Known prior leg fractures, patient has already undergone fasciotomy of the injured leg prior to enrollment
* History of peripheral vascular disease or concurrent lower extremity vascular injury/surgery
* Admission for atraumatic medical reasons
* Subject is unable to provide informed consent, or consent cannot be obtained from a legally authorized representative
* Complete spinal cord injuries, bilateral upper extremity injuries, or amputation/mangled lower extremity
* Patients who are in police custody at presentation to the hospital or who are pregnant
* Patient has an open injury on the injured leg that is large enough that at least one NIRS sensor cannot be safely placed over the compartment
* Bilateral leg injuries
* Not able to be enrolled within 48 hours after injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the trauma bay, surgical wards and ICU of Grady Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-07-20 (Actual); Study Completion 2016-07-20 (Actual)

PRIMARY OUTCOMES:
NIRS measurements as compared to clinical findings | Participants will be followed for the duration of hospital stay, an expected average of 72 hours
  Assess the accuracy of the Nonin 7600 oximeter with the Sensor Model 8004CV in the diagnosis of Acute Compartment Syndrome, using the "gold standard" criterion for ACS, which will be "clinical diagnosis". That is, all subjects undergoing fasciotomy for clinically diagnosed ACS will be considered to have ACS. NIRS values will be compared to clinical diagnosis to determine accuracy and threshold values.

SECONDARY OUTCOMES:
Accuracy of NIRS measurements compared to Intracompartmental pressure (ICP) measurements | Participants will be followed for the duration of hospital stay, an expected average of 72 hours
  ICP measurements will be compared to NIRS values to assess the magnitude of accuracy between the 2 tools.
Correlation between NIRS measurements between injured and uninjured extremity | Participants will be followed for the duration of hospital stay, an expected average of 72 hours
  Compare NIRS values between non-injured and injured extremities

CONTACTS AND LOCATIONS:
Overall Officials: William Reisman, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States